CLINICAL TRIAL: NCT06663644
Title: Comparative Effectiveness of Muscle Energy Technique on Iliotibial Band Versus Hamstring and Abdominal Muscles Activation in Patients With Nonspecific Low Back Pain
Brief Title: Muscle Energy Technique in Patients With Nonspecific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01993 FareehaZehra
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Nonspecific Low Back Pain
Keywords: nonspecific low back pain; muscle energy technique; hamstring and abdominal muscle activation; 90/90 hip lift with balloon

STUDY DESIGN:
Intervention Model Description: The two treatment groups are muscle energy technique group and hamstring and abdominal muscle activation group. Patients in the muscle energy technique group will receive muscle energy technique on iliotibial band along with conventional treatment. In this technique, after positioning the patient was asked to apply 30% force against therapist force and hold that contraction for 7-10seconds and after that relax for 5seconds and when patient exhale. Therapists take muscle to new restriction barrier; hold this position for 10-60 seconds with 3-5 repetition. The other group will receive 90/90 hip lift with balloon. The technique is performed in supine lying position such that lie on back with feet on a wall and knees and hips bent at 90 degrees angle. Place a 4-6" ball between knees. Place right arm above head and a balloon in left hand. Now inhale through nose and slowly blow out into the balloon. Pause 3 seconds with tongue on the roof of mouth to prevent airflow out of the balloon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique (Active Comparator): Post isometric relaxation technique is performed after positioning the patient and was asked to apply 30% force against therapist force and hold that contraction for 7- 10seconds and after that relax for 5seconds and when patient exhale. Therapists take muscle to new restriction barrier; hold this position for 10-60 seconds . Technique is performed 3-5 reps along with conventional treatment for 3 consecutive weeks.
  Interventions: Other: Muscle energy technique on iliotibial band
- Hamstring and abdominal muscle activation (Experimental): Techniques which target hamstring and abdominal muscle activation is 90/90 hip lift with balloon. It is performed in supine lying position such that lie on back with feet on a wall and knees and hips bent at 90 degrees angle. Place a 4-6" ball between knees. Place right arm above head and a balloon in left hand. Now inhale through nose and slowly blow out into the balloon. Pause 3 seconds with tongue on the roof of mouth to prevent airflow out of the balloon. Slowly blow out as stabilize the balloon .it is performed along with conventional therapy of moist pack for 15 mins, pelvic bridging, pelvic rolling.
  Interventions: Other: Hamstring and abdominal muscle activation

INTERVENTIONS:
Other: Muscle energy technique on iliotibial band — Post isometric relaxation involves the peripheral and central modulating mechanism by activating the muscles and joint mechanoreceptors. It can be effective for a variety of purposes including lengthening a shortened muscles, as a lymphatic or venous pump to aid the drainage of fluid or blood and increasing the range of motion. MET is a manual therapy intervention that can be used to stretch or lengthen muscles and fascia that lack flexibility.
  Arms: Muscle energy technique
Other: Hamstring and abdominal muscle activation — The 90/90 exercises for abdominal and hamstring activation rotate the pelvis posteriorly in the sagittal and transverse plane, into a more neutral position. Hamstrings extend the hip, and therefore reciprocally inhibit hip flexors. Hamstrings and abdominals also aid in inhibiting paraspinal muscles via a posterior pelvic tilt / hip extension, a decrease in lumbar extension, and an increase in lumbar flexion.
  Arms: Hamstring and abdominal muscle activation

SUMMARY:
The aim of this Randomized control trial is to find out the comparative effects of muscle energy technique on iliotibial band versus hamstring and abdominal muscle activation in patients with non specific low back pain in improving pain intensity and functional disability. The sample size was 28. Subjects are randomly divided into two groups. 14 subjects in muscle energy technique group and 14 in hamstring and abdominal muscle activation group. Study duration was of 6 months. Sampling technique applied was Non probability purposive sampling. Subjects between the age group 18- 40 years with acute non specific low back were included. Tools used are Numeric pain rating scale and Oswestry disability index.

DETAILED DESCRIPTION:
Non-specific low back pain is a mechanical pain of musculoskeletal origin in which symptoms vary with the nature of physical activities. It manifests as pain, muscle tension, or stiffness that is localized below the costal margin and above the inferior gluteal folds and is not attributed to a specific pathology with or without leg pain involvement. The lower back area, which extends from the end of the ribs to the start of the legs, feels tight, painful, and rigid.

A study conducted to investigate the immediate effects of MET of Quadratus Lamborum in chronic low back pain patients with functional leg length discrepancy. The outcomes of the study concluded that MET showed significant changes in pelvic alignment, leg length, pain, and fatigue. In a research conducted in 2020 to see the effectiveness of exercise with balloon and interferential therapy for pain and disability in low back pain in young adults . This study concluded that greater effect of 90/90 bridge with ball and balloon exercise on patients with mechanical low back pain. Individuals with low back pain often exhibit reduced hamstring muscle flexibility and altered pelvic range of motion as shortened and inflexible hamstring muscles can exert tension on the pelvis, leading to non-specific low back pain and disruptions in lumbar pelvic rhythm. Addressing hamstring flexibility is crucial for effective management of low back pain. Moreover, disturbances in the lower extremity kinematic chain, particularly involving the iliotibial band (ITB), can further impact pelvic biomechanics. Poor muscle coordination and decreased intrinsic postural muscle activity may compromise spinal stability in individuals with low back pain. The rationale of the present study is to find out the effectiveness of muscle energy technique on iliotibial band versus hamstring and abdominal muscles activation in non-specific low back pain patients, pain and disability. To compare the effectiveness of muscle energy technique on iliotibial band and hamstring and abdominal muscles activation in non-specific low back pain patients in improving pain intensity and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age between 18 to 40 years.
* Participants with acute non specific low back pain.
* Participants with postural low back pain.

Exclusion Criteria:

* Participants of age more than 40 years.
* Patients with history of lumbopelvic surgery.
* Having history of spinal or pelvic fracture, trauma of motor vehicle accident, fracture of lower extremity.
* Participants having systemic disease such as arthritis, TB, liver or kidney failure.
* Participants suffering from osteoporosis, psychiatric disorders, hematomas or abscesses.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 3 weeks
  It is an 11-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicate the "worst imaginable pain". Patients are instructed to choose a single number from the scale that best indicates their level of pain.
Modified Oswestry disability index | 3 weeks
  It is one of the most common patient-reported outcome measures used to evaluate the impact of back pain on patients" activities of daily living. It is used to access pain-related disability in people with acute, sub acute, or chronic low back pain. It consists of 10 items- 1 item on pain while the other 9 items are on activities of daily living. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Shamaila Yaqub, Principal Investigator — Riphah International University
Locations (1):
- PHQ hospital Gilgit, Gilgit, Gilgit-Baltistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore SD, Laudner KG, McLoda TA, Shaffer MA. The immediate effects of muscle energy technique on posterior shoulder tightness: a randomized controlled trial. J Orthop Sports Phys Ther. 2011 Jun;41(6):400-7. doi: 10.2519/jospt.2011.3292. Epub 2011 Apr 6. PMID 21471651
- [Background] Tenney HR, Boyle KL, Debord A. Influence of Hamstring and Abdominal Muscle Activation on a Positive Ober's Test in People with Lumbopelvic Pain. Physiother Can. 2013 Winter;65(1):4-11. doi: 10.3138/ptc.2011-33. PMID 24381375
- [Background] Boyle KL, Demske JR. Management of a female with chronic sciatica and low back pain: a case report. Physiother Theory Pract. 2009 Jan-Feb;25(1):44-54. doi: 10.1080/09593980802622677. PMID 19140082
- [Background] Suresh A, Kashyap D, Behera TP, kumar Tarsolia A. Effect of Muscle Energy Technique in Patients with Non-traumatic Lumbo-pelvic Pain in the Age Group of 30-40 Years. Journal of Physical Medicine Rehabilitation Studies & Reports SRC/JPMRS/138. 2021:3
- [Background] Iizuka Y, Iizuka H, Mieda T, Tsunoda D, Sasaki T, Tajika T, Yamamoto A, Takagishi K. Prevalence of Chronic Nonspecific Low Back Pain and Its Associated Factors among Middle-Aged and Elderly People: An Analysis Based on Data from a Musculoskeletal Examination in Japan. Asian Spine J. 2017 Dec;11(6):989-997. doi: 10.4184/asj.2017.11.6.989. Epub 2017 Dec 7. PMID 29279756
- [Background] Franke H, Fryer G, Ostelo RW, Kamper SJ. Muscle energy technique for non-specific low-back pain. Cochrane Database Syst Rev. 2015 Feb 27;2015(2):CD009852. doi: 10.1002/14651858.CD009852.pub2. PMID 25723574
- [Background] Deshmukh M, Pokle S, Baxi G, Palekar T, Gopiyani I. The Effect of Quadratus Lumborum Muscle Energy Technique on Low Back Pain and Diaphragmatic Electrophysiological Outcomes. Iranian Rehabilitation Journal. 2023;21(4):695-702.
- [Background] Ellythy MA. Efficacy of muscle energy technique versus strain counter strain on low back dysfunction. Bull Fac Phys Ther. 2012;17(2):29-35.
- [Background] Yoon JD, Jung JH, Cho HY, Shin HJ. The Immediate Effects of Muscle Energy Technique in Chronic Low Back Pain Patients with Functional Leg Length Discrepancy: A Randomized and Placebo-Controlled Trial. Healthcare (Basel). 2023 Dec 26;12(1):53. doi: 10.3390/healthcare12010053. PMID 38200959
- [Background] Shetty CB, Fathima N. Effectiveness of Exercise with Balloon for Low Back Pain in Young Adults: A quasi experimental study. Indian Journal of Physiotherapy & Occupational Therapy Print-(ISSN 0973-5666) and Electronic-(ISSN 0973-5674). 2020;14(4):20-6.
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Smeets R, Koke A, Lin CW, Ferreira M, Demoulin C. Measures of function in low back pain/disorders: Low Back Pain Rating Scale (LBPRS), Oswestry Disability Index (ODI), Progressive Isoinertial Lifting Evaluation (PILE), Quebec Back Pain Disability Scale (QBPDS), and Roland-Morris Disability Questionnaire (RDQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S158-73. doi: 10.1002/acr.20542. No abstract available. PMID 22588742
- [Background] Mehra A, Baker D, Disney S, Pynsent PB. Oswestry Disability Index scoring made easy. Ann R Coll Surg Engl. 2008 Sep;90(6):497-9. doi: 10.1308/003588408X300984. Epub 2008 Jul 2. PMID 18598595
- [Background] Rishi P, Arora B. Impact of muscle energy technique along with supervised. Exercise program over muscle energy technique on quadratus lumborum and iliopsoas on pain and functional disability in chronic non specific low back pain. International Journal of Physiotherapy and Research. 2018;6(3):2748-53.
- [Background] . Sharma D, Sen S. Effects of muscle energy technique on pain and disability in subjects with SI joint dysfunction. Int J Physiother Res. 2014;2(1):305-11
- [Background] Cook CE, Garcia AN, Wright A, Shaffrey C, Gottfried O. Measurement Properties of the Oswestry Disability Index in Recipients of Lumbar Spine Surgery. Spine (Phila Pa 1976). 2021 Jan 15;46(2):E118-E125. doi: 10.1097/BRS.0000000000003732. PMID 33038201
- [Background] Kumar N, Kumar M, Chhabra C, Kaur H. Unveiling the Link between Pelvic Inclination and Hamstring Tightness in Middle-Aged Individuals Afflicted with Non-Specific Low Back Pain. Journal of the Dow University of Health Sciences (JDUHS). 2023;17(3).
- [Background] Kato S, Murakami H, Demura S, Yoshioka K, Shinmura K, Yokogawa N, Igarashi T, Yonezawa N, Shimizu T, Tsuchiya H. Abdominal trunk muscle weakness and its association with chronic low back pain and risk of falling in older women. BMC Musculoskelet Disord. 2019 Jun 3;20(1):273. doi: 10.1186/s12891-019-2655-4. PMID 31159812
- [Background] Ahmed UA, Maharaj SS, Van Oosterwijck J. Effects of dynamic stabilization exercises and muscle energy technique on selected biopsychosocial outcomes for patients with chronic non-specific low back pain: a double-blind randomized controlled trial. Scand J Pain. 2021 Feb 24;21(3):495-511. doi: 10.1515/sjpain-2020-0133. Print 2021 Jul 27. PMID 33641272
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187